CLINICAL TRIAL: NCT00678613
Title: Role of Probiotics in the Prevention of Spontaneous Bacterial Peritonitis in Cirrhotic Patients: A Randomized Placebo Control Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: SBP-Probiotics rct
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Spontaneous Bacterial Peritonitis; Liver Cirrhosis
Keywords: probiotics; cirrhosis; prophylaxis; cirrhotic; patients; with; ascites; using
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Ascites | interventions — Probiotics; Norfloxacin

ARMS (2):
- 1, Primary prophylaxis (Placebo Comparator): Patients with liver cirrhosis with ascites having ascitic fluid protein <1 gm/dl will be included in this arm.
  They will be randomized between probiotics and placebo.
  Interventions: Drug: Probiotics and Placebo
- 2, secondary prophylaxis (Active Comparator): Patients with liver cirrhosis with ascites having history of prior SBP will be included in this arm.
  They will be randomized between probiotics and norfloxacin.
  Interventions: Drug: Probiotics and Norfloxacin

INTERVENTIONS:
Drug: Probiotics and Placebo — The Probiotics used in this study will be VSL#3. The control will be given similar looking capsules containing galactose powder. It will be used in the form of capsules. A total dose of 450 billions CFU will be used. Norfloxacin, 400 mg /day, will also be used as similar looking capsules. The drugs and placebo will be given for one year or till the end points of the study.
  Arms: 1, Primary prophylaxis
Drug: Probiotics and Norfloxacin — The Probiotics used in this study will be VSL#3. The control will be given similar looking capsules containing galactose powder.It will be used in the form of capsules. A total dose of 450 billions CFU will be used. Norfloxacin, 400 mg /day, will also be used as similar looking capsules. The drugs will be given for one year or till the end points of the study.
  Arms: 2, secondary prophylaxis

SUMMARY:
Cirrhotic patients are predisposed to bacterial infection. A large proportion of which is spontaneous bacterial peritonitis(SBP), which are mainly caused by enteric bacteria.SBP in a cirrhotic patients is associated with a high mortality rate in the order of 30-80% per year.It has been demonstrated that cirrhotics who have an ascitic fluid protein concentration less than 1gm% are most susceptible to develop SBP by virtue of having low opsonising activity of ascitic fluid.Patients with liver cirrhosis have significant degrees of imbalance of intestinal flora.Translocation of intestinal bacteria being the major mechanism for the production of SBP.

Long-term antibiotic (norfloxacin) is very effective in preventing SBP caused by gram negative bacteria.But the problem with the long-term antibiotic prophylaxis is the potential for the development of infection with antibiotic-resistant bacteria.Further, quinolones have no effect on gram positive bacteria which is becoming one of the important cause of SBP.

Such experiences necessitate the need for strategies, other than antibiotic, to prevent intestinal bacterial overgrowth, bacterial translocation and SBP in patients with cirrhosis.Probiotics have been used successfully to alter the gut flora in many clinical conditions where growth and localization of non pathogenic bacteria replaces the pathogenic bacteria in the intestine.The probiotic bacteria, among which the most common are the lactose fermenting Lactobacilli, inhibit the growth of pathogenic bacteria by acidifying the gut lumen, competing for nutrients, and by producing antimicrobial substances. They adhere to the gut mucosa and by that are thought to prevent bacterial translocation from the gut.

The purpose of this study is to determine the effectiveness of probiotics in the prevention of spontaneous bacterial peritonitis in patients with cirrhosis with low protein ascites and those already have developed an episode SBP.

DETAILED DESCRIPTION:
AIMS :

To study the effect of a Probiotics administration in reducing the incidence of first episode of SBP among cirrhotics who have low protein(<1 gm/dl) ascites.

To study the effect of a Probiotics administration in reducing the incidence of second episode of SBP among cirrhotic who have already developed at least one episode of SBP.

Study design : Prospective randomized placebo control efficacy study.

Inclusion criteria: All patients with liver cirrhosis with ascites having either history of prior SBP or ascitic fluid protein <1 gm/dl will be included in the study irrespective of etiology.

Exclusion criteria :

* Patients chronically treated with antibiotics or lactulose during past 30 days.
* Patients having risk factor of small intestinal bacterial overgrowth other than cirrhosis - diabetes mellitus, history of abdominal surgery, immunomodulator drugs. Alcoholic cirrhotics who continue to take alcohol.
* Patients with active or recent G.I. bleed (within prior 7 days).
* Patients with advanced HCC, renal failure and portal vein thrombosis

Patients in primary prophylaxis group will be randomly allocated to receive either a Probiotics or placebo. While patients in secondary prophylaxis group will be randomized between Probiotics and norfloxacin.

The Probiotics used in this study will be VSL#3. The control will be given similar looking capsules containing galactose powder.It will be used in the form of capsules. A total dose of 450 billions CFU will be used. Norfloxacin will also be used as similar looking capsules. The drugs and placebo will be given for one year or till the end points of the study as mentioned below.

Monitoring Each patients will be tested for SBP( Ascitic fluid cell count as well as culture) at the interval of every 6 weeks till the end point of the study.The effect of Probiotics on gut flora will be assessed objectively by jejunal fluid culture analysis baseline at 6 months and 1 year of the start of the treatment. This will be done on some of the representative sample from both the groups. Development of an episode of SBP, hepatic encephalopathy and variceal bleeding will be noted.All patients will be prospectively followed up from the date of enrollment to see the primary outcome that is development of SBP. The secondary outcome of the study will be the development of encephalopathy, variceal bleeding ,renal failure and death of the patients.

End Points :

1. completion of one year.
2. development of an episode of SBP.
3. Death.

ELIGIBILITY:
Inclusion Criteria:

* All patients with liver cirrhosis with ascites having either history of prior SBP or ascitic fluid protein <1 gm/dl will be included in the study irrespective of etiology.

Exclusion Criteria:

* Patients chronically treated with antibiotics(that disturb/alter normal gut flora) or lactulose during past 30 days.
* Patients having risk factor of small intestinal bacterial overgrowth other than cirrhosis - diabetes mellitus, history of abdominal surgery, immunomodulator drugs. Alcoholic cirrhotics who continue to take alcohol.
* Patients with active or recent G.I. bleed (within prior 7 days).
* Patients with advanced HCC, renal failure and portal vein thrombosis.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-07

PRIMARY OUTCOMES:
Development of an episode of SBP, completion of one year, or death | till end points

SECONDARY OUTCOMES:
development of encephalopathy, variceal bleeding and renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Subrat K Acharya, DM, Principal Investigator — All India Institute of Medical Sciences, New Delhi, India
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Riordan SM, Williams R. The intestinal flora and bacterial infection in cirrhosis. J Hepatol. 2006 Nov;45(5):744-57. doi: 10.1016/j.jhep.2006.08.001. Epub 2006 Sep 1. No abstract available. PMID 16979776
- [Background] Wiest R, Garcia-Tsao G. Bacterial translocation (BT) in cirrhosis. Hepatology. 2005 Mar;41(3):422-33. doi: 10.1002/hep.20632. PMID 15723320
- [Background] Chiva M, Soriano G, Rochat I, Peralta C, Rochat F, Llovet T, Mirelis B, Schiffrin EJ, Guarner C, Balanzo J. Effect of Lactobacillus johnsonii La1 and antioxidants on intestinal flora and bacterial translocation in rats with experimental cirrhosis. J Hepatol. 2002 Oct;37(4):456-62. doi: 10.1016/s0168-8278(02)00142-3. PMID 12217598
- [Background] Liu Q, Duan ZP, Ha DK, Bengmark S, Kurtovic J, Riordan SM. Synbiotic modulation of gut flora: effect on minimal hepatic encephalopathy in patients with cirrhosis. Hepatology. 2004 May;39(5):1441-9. doi: 10.1002/hep.20194. PMID 15122774
- [Background] Rayes N, Seehofer D, Hansen S, Boucsein K, Muller AR, Serke S, Bengmark S, Neuhaus P. Early enteral supply of lactobacillus and fiber versus selective bowel decontamination: a controlled trial in liver transplant recipients. Transplantation. 2002 Jul 15;74(1):123-7. doi: 10.1097/00007890-200207150-00021. PMID 12134110